CLINICAL TRIAL: NCT02432911
Title: A Multicenter，Open-label，Randomized Study on the Treatment of Elderly Chinese Acute Myeloid Leukemia Patients Aged 65 to 75 Years Old
Brief Title: Treatment of Elderly Chinese Acute Myeloid Leukemia Patients Aged 65 to 75 Years Old
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianxiang Wang (Unknown)
Responsible Party: Sponsor-Investigator, Jianxiang Wang, vice-president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHBDH-IIT2015003
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CAG protocol; aclacinomycins; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAG regimen (Experimental): Aclacinomycin 20mg/d for 4 days combined with cytarabine 20mg bid for 10 days with/without G-CSF 6ug/m2 from 1 day before therapy to day 10 of therapy.
  Interventions: Drug: CAG regimen (Aclacinomycin, cytarabine, with/w/o G-CSF)
- Low dose cytarabine (Active Comparator): cytarabine 20mg bid for 10 days.
  Interventions: Drug: low dose cytarabine

INTERVENTIONS:
Drug: CAG regimen (Aclacinomycin, cytarabine, with/w/o G-CSF) — Aclacinomycin 20mg/d for 4 days combined with cytarabine 20mg bid for 10 days with/without G-CSF 6ug/m2 from 1 day before therapy to day 10 of therapy.
  Arms: CAG regimen
Drug: low dose cytarabine — cytarabine 20mg bid for 10 days.
  Other Names: cytarabine
  Arms: Low dose cytarabine

SUMMARY:
This study focus on the comparison of CAG regimen to the low dose cytarabine therapy in elderly AML patients who are unfit or unwilling to receive intensive chemotherapy.

DETAILED DESCRIPTION:
Low dose cytarabine remains to be the choice of standard for elderly AML patients who are unfit or unwilling to receive intensive treatment. CAG regimen, which is a combination of aclacinomycin，low dose cytarabine±G-CSF is used often in elderly AML patients in China. It is proved effective and safety in some pilot studies，while there is no prospective，randomized study yet.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia except APL
* ECOG PS：0-3
* Unfit or unwilling to receive intensive therapy

Exclusion Criteria:

* The one who has already received induction therapy no matter what the outcome is.
* Active cancer patients who are needed to receive treatment;
* Serious uncontrolled infectious diseases(eg.tuberculosis or invasive pulmonary aspergillosis）；
* Active heart disease

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
complete remission rate | 4 months
relapse free survival | 3 years
treatment-related mortality | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Treatment and Diagnosis Center of Leukemia, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided